CLINICAL TRIAL: NCT06458062
Title: Development and Validation of an Artificial-Intelligence-enabled Portable Colposcopy Device for Optimizing Triage Alternatives for HPV-based Cervical Cancer Screening
Brief Title: Pocket Colposcopy Using CARE Algorithm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Kenya Medical Research Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00114753; 1U01CA269192 (NIH)
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancer; HPV Infection
Keywords: HPV testing; colposcopy; cervical cancer screening
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Pocket Assisted Colposcopy (Experimental): Pocket-Assisted Visual Inspection with Acetic Acid (PA-VIA): The cervix should be wiped with a cotton swab to remove any preexisting mucous and/or blood. A 3-5% acetic acid solution will be applied using a spray bottle or fox swab. After approximately 1-minute, using the Pocket Colposcope any changes to the cervix will be noted. Using the Calla Health image acquisition software, both white and green images of the cervix will be captured at low-resolution. Acetic acid may be reapplied between white and green imaging at the provider's discretion if acetowhitening diminishes. Images will be acquired. A biopsy will be obtained using the pocket. Random biopsies will be obtained from 2 quadrants in the absence of a visible lesion.
  Interventions: Device: Pocket Colposcope

INTERVENTIONS:
Device: Pocket Colposcope — Each patient will receive treatment in order to prevent cervical cancer

SUMMARY:
The Pocket colposcope has 510k FDA clearance and has been successfully used in ~2500 unique patients globally in Duke and non-Duke protocols to date. 1054 women who are HPV(+) and planned to undergo treatment at four Ministry of Health-supported outpatient clinics in Kisumu County will be recruited to the study. After providing informed consent, participants will be proceed with colposcopy using the POCKET colposcope.

DETAILED DESCRIPTION:
Women undergo Pocket-Assisted VIA (PA-VIA) and green light imaging using the Pocket Colposcope. Women will have biopsies taken of any suspicious lesions, or two biopsies taken in random locations if no lesions are visible. The locations of the biopsies will be based on provider impression. After their study-exams and biopsies are taken, women who are eligible for ablative treatment will be immediately treated in the clinic. Those with larger lesions or lesions concerning for invasive cancer will be referred to the local hospital for an excisional procedure. Once we have obtained enough images to develop the CARE algorithm, it will also be used to assist the provider in diagnosis.

This record previously reflected only Phase 1 of Aim 3 of the grant. Phase 1 of Aim 3 was originally included within NCT04998318. The details for Phase 2 of Aim 3 were added to this record in September 2025 after approval.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 30 years old and ≤ 64 years old; or Age ≥ 25 years old if women living with HIV (WLWH)
2. Sex: Female
3. Positive HPV test within past 6 months

Exclusion Criteria:

1. Pregnant women (cannot perform a cervical biopsy on a patient who is pregnant unless absolutely indicated)
2. Women with a negative HPV test within the past 9 months
3. Patients incapable of giving informed consent
4. Women with a history of cervical cancer
5. Pelvic exam concerning for cervical cancer or cervical infection
6. History of hysterectomy

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1079 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the Pocket CARE in detecting pre-cancer | Day of imaging (Day 1)
  Sensitivity will be reported as a percentage
Specificity of the Pocket CARE in detecting pre-cancer | Day of imaging (Day 1)
  Specificity will be reported as a percentage
Positive Predictive Value (PPV) of the Pocket CARE in detecting pre-cancer | Day of imaging (Day 1)
  PPV will be reported as a percentage
Negative Predictive Value (NPV) of the Pocket CARE in detecting pre-cancer | Day of imaging (Day 1)
  NPV will be reported as a percentage

CONTACTS AND LOCATIONS:
Overall Officials: Megan Huchko, MD, Principal Investigator — Duke University
Locations (1):
- Kenya Medical Research Institute, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: No